CLINICAL TRIAL: NCT03785301
Title: Effect of FGM on Glucose Control in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KY20170904-04
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FGM group (Experimental): Diabetic patients will use FreeStyle Libre Flash Glucose Monitoring (FGM) system(unmasked) to monitor glucose level once a month for 3 months.
  Interventions: Device: Freestyle Libre Flash Glucose Monitoring
- SMBG group (No Intervention): Diabetic patients will use Standard Blood Glucose Monitoring (SMBG) to monitor glucose level for 3 months. A 14-day masked wear of FreeStyle Libre H Flash Glucose Monitoring system is included for these subjects once a month, to collect glycaemic variability data for comparison to the intervention group of the study.

INTERVENTIONS:
Device: Freestyle Libre Flash Glucose Monitoring — Freestyle Libre Flash Glucose Monitoring will be used in diabetic patients once a month for therr months to monitor glucose level. Patients could scan the sensor to get the glucose level at any time as they want. They could alter thier diet and exercise according to the glucose levels. Patients will be required to keep track of food and exercise during wearing FGM sensor. Physicians would adjust patients' medication according their glucose profile provided by FGM, A1c, and diet and exercise every month.
  Arms: FGM group

SUMMARY:
The aim of the study is to assess the eﬀect of FGM on glycemic control compared with SMBG using a randomised controlled study design in adults with type 2 diabetes.

DETAILED DESCRIPTION:
Flash glucose monitoring (FGM) is a newly introduced Glucose Monitoring system. The aim of the study is to assess the eﬀect of FGM on glycemic control compared with standard blood glucose monitoring (SMBG) using a randomised controlled study design in adults with type 2 diabetes. Subjects will use unmasked FGM once a month or SMBG to monitor glucose level for 3 months. Patients in the SMBG group will wear masked FGM to collect glycaemic variability data for comparison to the intervention group of the study. The primary outcome, HbA1c, will be cpmpared at baseline and 3 month. Glucose control parameters provided by unmasked and masked FGM will be compared in the two groups, including mean blood glucose (MBG), coefficient of variation (CV), area under the curve (AUC), Time in Range(TIR), etc.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old;
2. diagnosed as having diabetes who were willing to perform the study and complete the data collection;
3. in stable condition prior to the study.

Exclusion Criteria:

1. pregnancy or attempting to conceive;
2. known allergy to medical grade adhesive or isopropyl alcohol used to prepare the skin;
3. skin lesions, scarring, redness, infection, or edema at the sensor application sites;
4. patients whose conditions were extremely severe and not stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 3 months
  Difference in HbA1c between intervention and control group at 3 month adjusting for baseline HbA1c

SECONDARY OUTCOMES:
mean blood glucose (MBG) | 1,2,3 months
  Difference in HbA1c between intervention and control group at 1, 2, and 3 month.
coefficient of variation (CV) | 1,2,3 months
  Difference in CV between intervention and control group at 1, 2, and 3 month.
area under the curve (AUC)<3.9mmol/L and >10mmol/L | 1,2,3 months
  Difference in AUC<3.9mmol/L and >10mmol/L between intervention and control group at 1, 2, and 3 month.
Time in Range (TIR) | 1,2,3 months
  Difference in time in range 3.9-10 mmol/L between intervention and control group at 1, 2, and 3 month.
FGM accuracy | during FGM
  Accuracy of FGM values versus reference blood glucose values (Consensus Error Grid (CEG) analysis and calculation of the Mean Absolute Relative Difference (MARD)

CONTACTS AND LOCATIONS:
Overall Officials: Ma Jianhua, MD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hostital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Chen M, Li H, Shen Y, Liu B, Yan R, Sun X, Ye L, Lee KO, Ma J, Su X. Flash Glucose Monitoring Improves Glucose Control in People with Type 2 Diabetes Mellitus Receiving Anti-diabetic Drug Medication. Exp Clin Endocrinol Diabetes. 2021 Dec;129(12):857-863. doi: 10.1055/a-0994-9850. Epub 2020 Aug 28. PMID 32858752
- [Derived] Hu Y, Shen Y, Yan R, Li F, Ding B, Wang H, Su X, Ma J. Relationship Between Estimated Glycosylated Hemoglobin Using Flash Glucose Monitoring and Actual Measured Glycosylated Hemoglobin in a Chinese Population. Diabetes Ther. 2020 Sep;11(9):2019-2027. doi: 10.1007/s13300-020-00879-x. Epub 2020 Jul 21. PMID 32696267